CLINICAL TRIAL: NCT06541626
Title: Sun Yat-Sen Prospective Cohort Study of Central Nervous System Idiopathic Inflammatory Demyelinating Diseases
Brief Title: Sun Yat-Sen Cohort of CNS Idiopathic Inflammatory Demyelinating Diseases
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-109-01
Record Dates: First submitted 2024-07-11; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis, MS; Neuromyelitis Optica Spectrum Disorders; Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease; Acute Disseminated Encephalomyelitis; Clinically Isolated Syndrome; Demyelinating Disorder
Keywords: CNS IIDD; follow-up
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Encephalomyelitis, Acute Disseminated; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- MS: Diagnosis meets the 2017 McDonald diagnostic criteria, receive the recommended diagnosis and treatment plans from current international and national guidelines or expert consensus.
- NMOSD: Diagnosis meets the 2015 IPND diagnostic panel standards, receive the recommended diagnosis and treatment plans from current international and national guidelines or expert consensus.
- MOGAD: Diagnosis meets the 2023 international expert panel recommended standards, receive the recommended diagnosis and treatment plans from current international and national guidelines or expert consensus.
- ADEM: Diagnosis meets the diagnostic criteria for ADEM
- CIS: Diagnosis meets the 2017 McDonald diagnostic criteria, receive the recommended diagnosis and treatment plans from current international and national guidelines or expert consensus.
- undefined CNS IIDD: First occurrence of CNS inflammatory demyelinating event, not yet diagnosable as MS, NMOSD, MOGAD, ADEM, or other definitive types of central nervous system demyelinating diseases, with symptoms and signs lasting more than 24 hours

SUMMARY:
The goal of this observational study is to learn about pathogenesis and clinical prognosis of CNS IIDD in the Chinese population and to provide evidence-based clues for clinical treatment decisions.

The main questions it aims to answer are:

Question 1: Clarify the clinical characteristics and prognostic factors of various diseases (MS, NMOSD, MOGAD, etc.) within IIDD in the Chinese population.

Question 2: Analyze the relationship between biomarkers and the occurrence, progression, and prognosis of CNS IIDD cases in our hospital.

Participants will

1. Receive the recommended diagnosis and treatment plans from current international and national guidelines or expert consensus, without additional special interventions.
2. Receive clinical evaluation, follow-up, and management from dedicated neuroimmunology specialists.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65 years with central nervous system idiopathic inflammatory demyelinating diseases (CNS IIDD);
2. The clinical syndrome of the attack meets one of the following: MS, NMOSD, MOGAD, ADEM, clinically isolated syndrome, demyelinating encephalopathy, demyelinating myelitis, or brainstem encephalitis (see below A-E);
3. Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. History of tumors or diagnosis of central nervous system tumors;
2. Infectious lesions of the central nervous system;
3. Hereditary, metabolic, toxic, vascular, or traumatic demyelinating diseases of the brain/spinal cord;
4. Non-compliance with treatment and follow-up.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are aged between 18 and 65 years and diagnosed with central nervous system idiopathic inflammatory demyelinating diseases
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse | Through study completion, an average of 5 years
  Must meet the following criteria：① Appearance of new symptoms or worsening of existing symptoms;② Symptoms attributed to CNS IIDD;③ Duration ≥24 hours;④ Increase in clinical scores (e.g., EDSS);⑤ Imaging or electrophysiological tests clearly showing new responsible lesions.
Long-term neurological function | Through study completion, an average of 5 years
  Assessed using the Expanded Disability Status Scale (EDSS)，EDSS score ranges from 0 to 10, with 0 indicating a normal healthy state, 10 indicating death, and higher scores reflecting more severe disability.

SECONDARY OUTCOMES:
Long-term neurological function | Baseline, six months, one year, two years, and average three years
  Assessed using the Optic Spinal Impairment Scale (OSIS) and its sub-scores, OSIS score ranges from 0 to 25, and higher scores reflect more severe disability. OSIS sub-score ranges from 0 to 5-8, and higher scores reflect more severe in each component assessment.
Sub-scores of the Expanded Disability Status Scale (EDSS) | Baseline, six months, one year, two years, and average three years
  EDSS sub-score ranges from 0 to 5 or 6, with 0 indicating a normal healthy state, higher scores indicating worse neurological functions.
Optical coherence tomography (OCT) of the eyes: retinal nerve fiber layer thickness, macular thickness | Baseline, six months, one year, two years, and average three years
  The thickness is measured by machines by milimetres
Changes in humoral immune markers | Baseline, six months, one year, two years, and average three years
  The levels of neurofilament light chain (NfL), soluble GFAP, soluble TREM2, and other potential biomarkers are measured in g/ml.
Changes in pathogenic antibody titers | Baseline, six months, one year, two years, and average three years
  Titers of antibodies for MOG, AQP4, MBP, and AFO in iu/l
P100 amplitude of visual evoked potentials | Baseline, six months, one year, two years, and average three years
  Amplitude in volts
P100 latency of visual evoked potentials | Baseline, six months, one year, two years, and average three years
  Latency in seconds
Latency of somatosensory evoked potentials; | Baseline, six months, one year, two years, and average three years
  Latency in seconds
Latency of brainstem auditory evoked potentials; | Baseline, six months, one year, two years, and average three years
  Latency in seconds
Amplitude of somatosensory evoked potentials; | Baseline, six months, one year, two years, and average three years
  Amplitude in volts
Amplitude of brainstem auditory evoked potentials; | Baseline, six months, one year, two years, and average three years
  Amplitude in volts

OTHER OUTCOMES:
Recording of adverse reactions | Baseline, six months, one year, two years, and average three years
Follow-up of common adverse reactions | Baseline, six months, one year, two years, and average three years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No